CLINICAL TRIAL: NCT02043912
Title: Drug Interactions With Risk of QT-prolongation in a General Hospital: an Epidemiological Point Prevalence Study
Brief Title: Drug Interactions With Risk of QT-prolongation in a General Hospital
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Eline Vandael, PhD-student, KU Leuven
Other Study IDs: EV002
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: QT-prolongation
Keywords: QT-prolongation; Torsade de Pointes; Haloperidol; Drug interactions
MeSH Terms: conditions — Long QT Syndrome; Torsades de Pointes | interventions — Haloperidol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients treated with haloperidol
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Haloperidol
  Other Names: Haldol

SUMMARY:
In this epidemiological point prevalence study, medication profiles of patients with haloperidol treatment will be checked for drug interactions with risk of QT-prolongation. Additional clinical risk factors for developing QT-prolongation and safety measurements will be documented.

DETAILED DESCRIPTION:
Study design: epidemiological point prevalence study

Target population: Patients with haloperidol treatment

The following aspects will be investigated:

* The medication profiles will be checked for drug interactions with risk of QT-prolongation.
* Clinical risk factors for developing QT-prolongation (gender, age, (history of) cardiovascular disease, comorbidity,...) and lab results will be collected.
* Safety measurements (e.g. ECG) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* treatment with haloperidol (started in the hospital)

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are treated with haloperidol (every tuesday we will make a selection of the patients who received haloperidol on monday)
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
QTc-interval (corrected for heart rate) | maximum one year before inclusion / one week after inclusion

SECONDARY OUTCOMES:
number of drug interactions (with risk of QT-prolongation) | one week before/after inclusion

OTHER OUTCOMES:
number of patients with an ECG before or after the start of haloperidol | maximum one year before inclusion / one week after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Eline Vandael, PhD-student, Principal Investigator — KU Leuven
Locations (1):
- Universitair Ziekenhuis Leuven, Leuven, Belgium